CLINICAL TRIAL: NCT03009669
Title: The Application of Pleth Variability Index in Continuous Monitoring Volume Status in Patients Undergoing Intestinal Tumor Surgery
Brief Title: The Application of Pleth Variability Index in Continuous Monitoring the Volume Status of Intraoperative Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Guangzhou Panyu Central Hospital (Other)
Responsible Party: Principal Investigator, Lin Yang, attending physician, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: H20160049（01）
Record Dates: First submitted 2016-12-30; First posted 2017-01-04 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-12

CONDITIONS: Hemodynamic Monitoring
Keywords: pleth variability index; stroke volume variation; perfusion Index; intraoperative; intestinal tumor
MeSH Terms: conditions — Intestinal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To assess the value of using pleth variability index(PVI) to monitor the patient's intra-operative volume status continuously by observing the application of stroke volume variation(SVV) and PVI and their correlation in patients undergoing intestinal tumor surgeries.

DETAILED DESCRIPTION:
Objective: To assess the value of using PVI to monitor the patient's intra-operative volume status continuously by observing the application of stroke volume variation(SVV) and pleth variability index(PVI) and their correlation in patients undergoing intestinal tumor surgeries.

Methods: 50 patients undergoing elective intestinal tumor surgery were enrolled, ASAⅠ-Ⅲ, aged 18-65 years. After the induction of general anesthesia, cardiac index(CI), cardiac output(CO), stroke volume variability(SVV), stroke volume index(SVI) were monitored with Vigileo system, while pleth variability index(PVI) and perfusion index(PI) were monitored with Massion Radical 7 system. During the surgery, goal directed fluid therapy was conducted according to the data of CI、SVI and SVV. Heart rate(HR), mean arterial pressure(MAP), central venous pressure(CVP), CO, CI, SVI, SVV, PI, PVI were recorded while after the induction of anesthesia(T1), making surgical incision(T2), performing intestinal anastomosis(T3) and closing the abdominal incision(T4). And we calculate the correlation of SVV and PVI using Pearson Correlation Analysis at different time points.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective intestinal tumor surgery
* American Society of Anesthesiologists (ASA) physical status of grade I-Ⅲ
* Aged 18-65 years
* BMI 18~30kg/㎡

Exclusion Criteria:

* Patients under 18 years or above 65 years
* patients with severe aortic regurgitation
* patients with permanent cardiac arrhythmias
* patients with intra-aortic balloon pump
* patients with severe pulmonary disease
* patients undergoing emergency surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50 patients undergoing elective intestinal tumor surgery were enrolled, ASAⅠ-Ⅲ,aged 18-65 years,BMI 18~30kg/㎡.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-07 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
the correlation of SVV and PVI | during the surgery
  SVV and PVI were recorded while after the induction of anesthesia(T1),making surgical incision(T2),performing intestinal anastomosis(T3) and closing the abdominal incision(T4). We calculate the correlation of SVV and PVI using Pearson Correlation Analysis at different time points.

SECONDARY OUTCOMES:
stroke volume variability(SVV) | during the surgery
  stroke volume variability(SVV) in percentage.Record the date of SVV while after the induction of anesthesia(T1), making surgical incision(T2), performing intestinal anastomosis(T3) and closing the abdominal incision(T4).Compare the differences of SVV between the time points.
pleth variability index(PVI) | during the surgery
  pleth variability index(PVI) in percentage.Record the date of PVI while after the induction of anesthesia(T1), making surgical incision(T2), performing intestinal anastomosis(T3) and closing the abdominal incision(T4).Compare the differences of PVI between the time points.
pleth index(PI) | during the surgery
  pleth index(PI) in percentage.Record the date of PI while after the induction of anesthesia(T1), making surgical incision(T2), performing intestinal anastomosis(T3) and closing the abdominal incision(T4).Compare the differences of PI between the time points.
cardiac index(CI) | during the surgery
  cardiac index(CI) in L•min-1•m-2.Record the date of CI while after the induction of anesthesia(T1), making surgical incision(T2), performing intestinal anastomosis(T3) and closing the abdominal incision(T4).Compare the differences of CI between the time points.
stroke volume index(SVI) | during the surgery
  (SVI) in ml•m-2.Record the date of SVI while after the induction of anesthesia(T1), making surgical incision(T2), performing intestinal anastomosis(T3) and closing the abdominal incision(T4).Compare the differences of SVI between the time points.

CONTACTS AND LOCATIONS:
Overall Officials: Shu HaiHua, doctor, Study Chair — First Affiliated Hospital, Sun Yat-Sen University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Brandstrup B. Fluid therapy for the surgical patient. Best Pract Res Clin Anaesthesiol. 2006 Jun;20(2):265-83. doi: 10.1016/j.bpa.2005.10.007. PMID 16850777
- [Result] Grocott MPW, Mythen MG, Gan TJ. Perioperative fluid management and clinical outcomes in adults. Anesth Analg. 2005 Apr;100(4):1093-1106. doi: 10.1213/01.ANE.0000148691.33690.AC. PMID 15781528
- [Result] Nisanevich V, Felsenstein I, Almogy G, Weissman C, Einav S, Matot I. Effect of intraoperative fluid management on outcome after intraabdominal surgery. Anesthesiology. 2005 Jul;103(1):25-32. doi: 10.1097/00000542-200507000-00008. PMID 15983453
- [Result] Strunden MS, Heckel K, Goetz AE, Reuter DA. Perioperative fluid and volume management: physiological basis, tools and strategies. Ann Intensive Care. 2011 Mar 21;1(1):2. doi: 10.1186/2110-5820-1-2. PMID 21906324
- [Result] Samra T, Arya VK. Comparison of cardiac output estimation by FloTrac/Vigileo TM and intermittent pulmonary artery thermodilution in patient with Takayasu arteritis. Ann Card Anaesth. 2011 May-Aug;14(2):163-4. doi: 10.4103/0971-9784.81579. No abstract available. PMID 21636945
- [Result] Cannesson M. Arterial pressure variation and goal-directed fluid therapy. J Cardiothorac Vasc Anesth. 2010 Jun;24(3):487-97. doi: 10.1053/j.jvca.2009.10.008. No abstract available. PMID 20022261
- [Result] Mathews L, Singh RK. Cardiac output monitoring. Ann Card Anaesth. 2008 Jan-Jun;11(1):56-68. doi: 10.4103/0971-9784.38455. PMID 18182765
- [Result] Cannesson M, Attof Y, Rosamel P, Joseph P, Bastien O, Lehot JJ. Comparison of FloTrac cardiac output monitoring system in patients undergoing coronary artery bypass grafting with pulmonary artery cardiac output measurements. Eur J Anaesthesiol. 2007 Oct;24(10):832-9. doi: 10.1017/S0265021507001056. Epub 2007 Aug 1. PMID 17666154
- [Result] Rex S, Brose S, Metzelder S, Huneke R, Schalte G, Autschbach R, Rossaint R, Buhre W. Prediction of fluid responsiveness in patients during cardiac surgery. Br J Anaesth. 2004 Dec;93(6):782-8. doi: 10.1093/bja/aeh280. Epub 2004 Oct 1. PMID 15465840
- [Result] Michard F, Alaya S, Zarka V, Bahloul M, Richard C, Teboul JL. Global end-diastolic volume as an indicator of cardiac preload in patients with septic shock. Chest. 2003 Nov;124(5):1900-8. doi: 10.1378/chest.124.5.1900. PMID 14605066
- [Result] Mayer J, Boldt J, Mengistu AM, Rohm KD, Suttner S. Goal-directed intraoperative therapy based on autocalibrated arterial pressure waveform analysis reduces hospital stay in high-risk surgical patients: a randomized, controlled trial. Crit Care. 2010;14(1):R18. doi: 10.1186/cc8875. Epub 2010 Feb 15. PMID 20156348
- [Result] Haas S, Trepte C, Hinteregger M, Fahje R, Sill B, Herich L, Reuter DA. Prediction of volume responsiveness using pleth variability index in patients undergoing cardiac surgery after cardiopulmonary bypass. J Anesth. 2012 Oct;26(5):696-701. doi: 10.1007/s00540-012-1410-x. Epub 2012 May 16. PMID 22588287
- [Result] Zimmermann M, Feibicke T, Keyl C, Prasser C, Moritz S, Graf BM, Wiesenack C. Accuracy of stroke volume variation compared with pleth variability index to predict fluid responsiveness in mechanically ventilated patients undergoing major surgery. Eur J Anaesthesiol. 2010 Jun;27(6):555-61. doi: 10.1097/EJA.0b013e328335fbd1. PMID 20035228
- [Result] Desgranges FP, Desebbe O, Ghazouani A, Gilbert K, Keller G, Chiari P, Robin J, Bastien O, Lehot JJ, Cannesson M. Influence of the site of measurement on the ability of plethysmographic variability index to predict fluid responsiveness. Br J Anaesth. 2011 Sep;107(3):329-35. doi: 10.1093/bja/aer165. Epub 2011 Jun 16. PMID 21680600
- [Result] Monnet X, Teboul JL. Volume responsiveness. Curr Opin Crit Care. 2007 Oct;13(5):549-53. doi: 10.1097/MCC.0b013e3282ec68b2. PMID 17762234
- [Result] Sandroni C, Cavallaro F, Marano C, Falcone C, De Santis P, Antonelli M. Accuracy of plethysmographic indices as predictors of fluid responsiveness in mechanically ventilated adults: a systematic review and meta-analysis. Intensive Care Med. 2012 Sep;38(9):1429-37. doi: 10.1007/s00134-012-2621-1. Epub 2012 Jun 26. PMID 22732902
- [Result] Schoonjans A, Forget P, Labriola L, Deneys V, Jadoul M, Pingaut I, De Kock M. Pleth variability index combined with passive leg raising-induced pulse pressure variation to detect hypovolemia in spontaneously breathing patients. Acta Anaesthesiol Belg. 2010;61(3):147-50. PMID 21268570
- [Result] Takeyama M, Matsunaga A, Kakihana Y, Masuda M, Kuniyoshi T, Kanmura Y. Impact of skin incision on the pleth variability index. J Clin Monit Comput. 2011 Aug;25(4):215-21. doi: 10.1007/s10877-011-9298-9. Epub 2011 Sep 18. PMID 21928109